CLINICAL TRIAL: NCT01049282
Title: A Safety and Immunogenicity Phase 1 Trial With an Adjuvanted TB Subunit Vaccine (Ag85B-ESAT-6 + IC31) Administered in Different Antigen/Adjuvant Formulations in TST Negative and TST Positive Volunteers at 0 and 2 Months
Brief Title: A Safety and Immunogenicity Trial With an Adjuvanted TB Subunit Vaccine (Ag85B-ESAT-6 + IC31)
Acronym: THYB-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: THYB-03
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
Keywords: safety; immunogenicity; adjuvanted TB subunit vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 12 TST negative volunteers antigen only (Experimental)
  Interventions: Biological: Antigen (Ag85B-ESAT-6)
- 12 TST negative volunteers (Experimental)
  Interventions: Biological: Antigen (Ag85B-ESAT-6) with adjuvant (IC31)
- 12 BCG vaccinated volunteers (Experimental)
  Interventions: Biological: Antigen (Ag85B-ESAT-6) with adjuvant (IC31)
- 12 with Latent TB infection >= 2 years ago (Experimental)
  Interventions: Biological: Antigen (Ag85B-ESAT-6) with adjuvant (IC31)

INTERVENTIONS:
Biological: Antigen (Ag85B-ESAT-6) — Solution for injection, 0.5 mL, 50 ug antigen, 2 vaccinations with 2 months interval
  Arms: 12 TST negative volunteers antigen only
Biological: Antigen (Ag85B-ESAT-6) with adjuvant (IC31) — Suspension for injection, 0.5 mL, 50 ug antigen, 2 vaccinations with 2 months interval
  Arms: 12 BCG vaccinated volunteers; 12 TST negative volunteers; 12 with Latent TB infection >= 2 years ago

SUMMARY:
The study has the following objectives:

Primary objective To evaluate the safety profile of an adjuvanted TB subunit vaccine administered in different antigen/adjuvant formulations at 0 and 2 months Secondary objective To determine the immunogenicity profile of an adjuvanted TB subunit vaccine administered in different antigen/adjuvant formulations at 0 and 2 months.

DETAILED DESCRIPTION:
Number of trial subjects=48 Investigational product=Ag85B - ESAT-6 + IC31 Dosage Group 1: TST negative, 50 µg antigen Group 2: TST negative, 50 µg antigen + fixed adjuvant Group 3: BCG vaccinated, 50 µg antigen + fixed adjuvant Group 4 : Latent TB, 50 µg antigen + fixed adjuvant Dosage volume 0.5 ml Administration Intramuscularly into deltoid muscle, alternate arms at day 0 (right) and day 56 (left).

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 40 years old
* TST negative groups: TST- and negative QuantiFERON-TB Gold In tube test
* BCG group: known to be BCG-vaccinated > 2 years before(scar, vaccination card), TST+ (> 6 or any documented value > 6 mm on medical file in the past), with no active, chronic or past TB disease as confirmed by chest X ray, negative QuantiFERON-TB Gold In Tube test and negative 6-day lymphocyte tests.
* Infection group: latent TB, TST+ ( = or > 10 mm or documented = or > 10 mm positive on medical file in the past), previously TB infected but with no active disease confirmed by chest X ray, may have received chemoprophylaxis but with no TB treatment/chemoprophylaxis within the preceding 2 years, positive QuantiFERON-TB Gold In Tube test and/or positive 6-day lymphocyte test.
* Healthy based on medical examination/history at the inclusion
* Signed informed consent
* Prepared to grant authorized persons access to the medical records
* The volunteer is likely to comply with instructions

Exclusion Criteria:

* Confirmed active TB based on clinical evaluation(history, physical findings and investigations)
* Vaccinated with any vaccine 3 months before first vaccination
* Administration of immune modulating drugs (steroids, immunosuppressive drugs or immunoglobulins)
* HBV, HCV or HIV sero-positive
* Participation in other clinical trials
* Known hypersensitivity to any of the vaccine components
* Laboratory parameters outside of normal range considered clinically relevant

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety on Physical examination , and Laboratory safety tests of hematology clinical chemistry | 12 visits in a total of 224 days duratiion from the day of first vaccinantion

SECONDARY OUTCOMES:
Immunogenicity assessment by: A.Detection of IFN gama production after stimulation with Ag85B, ESAT-6 and H1. B.Detection of IgG antibodies to recombinant proteins Ag85B, ESAT-6 and H1 in serum/plasma. | 12 visits in a total of 224 days duratiion from the day of first vaccinantion

CONTACTS AND LOCATIONS:
Overall Officials: Jemal Hussein, MD, Principal Investigator — Armauer Hansen Research Institue/AHRI/,Ethiopia; Peter Bang, Msc, Study Director — Statens serum Institute/SSI/,Denamrk

REFERENCES:
- [Derived] Hussein J, Zewdie M, Yamuah L, Bedru A, Abebe M, Dagnew AF, Chanyalew M, Yohannes AG, Ahmed J, Engers H, Doherty TM, Bang P, Kromann I, Hoff ST, Aseffa A. A phase I, open-label trial on the safety and immunogenicity of the adjuvanted tuberculosis subunit vaccine H1/IC31(R) in people living in a TB-endemic area. Trials. 2018 Jan 10;19(1):24. doi: 10.1186/s13063-017-2354-0. PMID 29321075